CLINICAL TRIAL: NCT05473052
Title: Home-based Preoperative Exercise Training for Lung Cancer Patients Undergoing Surgery: A Feasibility Trial
Brief Title: Home-based Exercise Training for Lung Cancer Patients Awaiting Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Leiria (Other)
Responsible Party: Principal Investigator, Pedro Machado, Principal Investigator, Instituto Politécnico de Leiria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HomeFittosurgery
Record Dates: First submitted 2022-07-22; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Lung Neoplasm
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative home-based exercise training (Experimental): Patients received usual care plus a preoperative home-based exercise program consisting of aerobic and resistance exercise. In addition, a physical therapist carried out weekly telephone supervision with all participants
  Interventions: Behavioral: Preoperative home-based exercise training

INTERVENTIONS:
Behavioral: Preoperative home-based exercise training — 1) Home-based aerobic and resistance exercise training (preoperative period)
  Dose of aerobic exercise:
  1. Type: Walking
  2. Frequency: 3 sessions per week
  3. Duration: 30 minutes
  4. Intensity: Rate of perceived exertion on Borg Category Ratio-10 (3-5)
  5. Progression: Increase the walking duration in 10 minutes (after week 2)
  Dose of resistance exercise:
  1. Type: Six exercises for upper and lower limbs using bodyweight and free-wights of 1-2kg
  2. Frequency: 2 sessions per week
  3. Duration: 2 sets x 15 repetitions
  4. Rest in-between sets: 45 seconds
  5. Intensity:Rate of perceived exertion on Borg Category Ratio-10 (3-5)
  6. Progression: Increase the number of sets (3 sets of 15 repetitions after week
  2) Weekly telephone supervision: A physical therapist carried out weekly telephone calls with all participants to monitor adverse events, give positive reinforcement and recommend strategies to overcome barriers that arise during the exercise program.

SUMMARY:
Surgical resection is the only curative treatment in patients diagnosed with lung cancer, the most mortal type of malignancy globally. However, following lung cancer resection, patients experience a substantial deterioration in health-related quality of life and have an increased risk of developing pulmonary complications.

Although current clinical guidelines strongly recommend preoperative exercise training to improve clinical outcomes after lung cancer surgery, inaccessibility to facility-based exercise programs is a major barrier to routine participation, with patients indicating a strong preference to exercise in a home-based environment.

The primary purpose of the present study was to evaluate the feasibility of a home-based exercise program (HBEP) in lung cancer patients awaiting surgical treatment. The secondary purposes were to evaluate the safety of the HBEP and to explore exercise effects on patients' HRQOL and physical performance, either pre-and post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for surgical treatment of suspected or confirmed lung cancer (clinical stage IIIA or less)
* Waiting time for surgery of at least two weeks from baseline assessment
* Medical clearance to exercise.
* Signed informed consent prior to initiation of study-related procedures.

Exclusion Criteria:

* Metastatic cancer
* Presence of physical or mental disabilities that contraindicated exercise training or physical testing
* Unable to communicate in Portuguese or English
* Performing combined aerobic plus resistance training over the past month (self-reported ≥2 days a week, ≥30 minutes each session).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Baseline
  Defined as the ratio of recruited patients to those who were eligible, expressed as a percentage.
Retention rate | Baseline to 4-5 weeks after surgery
  Defined as the ratio of patients who completed the study to those who were recruited, expressed as a percentage
Exercise attendance rate | Baseline to 2-3 days before surgery
  Attendance rate will be defined as the ratio of total completed to planned exercise sessions, expressed as a percentage.
Exercise compliance rate | Baseline to 2-3 days before surgery
  Compliance rate will be defined as the ratio of total completed to planned training volume, expressed as a percentage.

SECONDARY OUTCOMES:
Adverse events | Baseline to 2-3 days before surgery
  Defined as any unfavorable or unexpected event that occurred as a direct result of exercise training, during or within 24 hours after an exercise session. The severity of adverse events was categorized based on the Common Terminology Criteria for Adverse Events (CTCAE), version 5. The CTCAE provides a grading (severity) scale, with each adverse event been classified as grade 1 (asymptomatic or mild symptoms, clinical or diagnostic observations only, and/or intervention not indicated) to grade 5 (death). An adverse event was classified as "serious" if it resulted in hospitalization, persistent or significant disability, was life threatening, or resulted in death (i.e., grade 3 or higher).
Changes in exercise capacity | Baseline to 2-3 days before surgery
  Assessed by the Incremental Shuttle Walk Test (ISWT). The ISWT measures the distance in meters an individual can walk around a 10 meters shuttle course paced according to an incremental speed dictated by an audio recording and was performed under the supervision of a single investigator using the protocol described by Singh et al.
  (1992). The test finished when the participant can no longer maintain the desired speed or became too breathless to continue.
Changes in exercise capacity | Baseline to 4-5 weeks after surgery.
  Assessed by the Incremental Shuttle Walk Test (ISWT). The ISWT measures the distance in meters an individual can walk around a 10 meters shuttle course paced according to an incremental speed dictated by an audio recording and was performed under the supervision of a single investigator using the protocol described by Singh et al.
  (1992). The test finished when the participant can no longer maintain the desired speed or became too breathless to continue.
Changes in health-related quality of life | Baseline to 2-3 days before surgery
  Assessed through the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire C30 (QLQ-C30) (version 3.0). The QLQ-C30 is composed of 30 questions, including five multi-item functioning scales, three multi-item symptom scales, six single-item symptom scales, and a two-item global health status scale [GHS]. Scores range from 0 to 100 points, with a higher score on the functioning scales indicating a higher level of functioning, whereas a higher score on the symptom scales indicates a higher level of symptom burden.
  In addition, was assessed the EORTC QLQ-C30 summary score (SumSc) because it provides a psychometrically more robust alternative to the GHS score that is frequently used as the primary HRQOL endpoint in clinical trials. The SumSc is calculated from the mean of 13 of the 15 QLQ-C30 scores (the GHS and financial impact scales are excluded).
Changes in health-related quality of life | Baseline to 4-5 weeks after surgery
  Assessed through the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire C30 (QLQ-C30) (version 3.0). The QLQ-C30 is composed of 30 questions, including five multi-item functioning scales, three multi-item symptom scales, six single-item symptom scales, and a two-item global health status scale [GHS]. Scores range from 0 to 100 points, with a higher score on the functioning scales indicating a higher level of functioning, whereas a higher score on the symptom scales indicates a higher level of symptom burden.
  In addition, was assessed the EORTC QLQ-C30 summary score (SumSc) because it provides a psychometrically more robust alternative to the GHS score that is frequently used as the primary HRQOL endpoint in clinical trials. The SumSc is calculated from the mean of 13 of the 15 QLQ-C30 scores (the GHS and financial impact scales are excluded).
Changes in handgrip strength | Baseline to 2-3 days before surgery
  Assessed using a Jamar hydraulic hand dynamometer (JA Preston Corporation, Jackson, MI, USA). Measurements were conducted using the standard position approved by the American Society of Hand Therapists. The standard adjustable handle dynamometer was set at the second handle position for all patients. The non-tested arm was resting neutrally and both feet were firmly on the ground, shoulder width apart. Patients were instructed to grip the handle with maximal strength during 3 seconds and the measurements were repeated three times for the left and right hand, with 30 seconds rest in-between measurements. The highest value for both hands (in kilograms) was considered as the output measure to each patient.
Changes in handgrip strength | Baseline to 4-5 weeks after surgery
  Assessed using a Jamar hydraulic hand dynamometer (JA Preston Corporation, Jackson, MI, USA). Measurements were conducted using the standard position approved by the American Society of Hand Therapists. The standard adjustable handle dynamometer was set at the second handle position for all patients. The non-tested arm was resting neutrally and both feet were firmly on the ground, shoulder width apart. Patients were instructed to grip the handle with maximal strength during 3 seconds and the measurements were repeated three times for the left and right hand, with 30 seconds rest in-between measurements. The highest value for both hands (in kilograms) was considered as the output measure to each patient.
Changes in five times sit to stand test | Baseline to 2-3 days before surgery
  Patients were instructed to perform the Five Times Sit to Stand Test (5STS) on a standardized armless chair (i.e., seating height between 41-45 cm, no elbow rests and wheels). After the cue "ready, set, go!", patients started the STS repetitions as rapidly as possible from the sitting position with their buttocks touching the chair to the full standing position, with their arms crossed over the chest. The 5STS test finished when the patients sit on the chair after the fifth repetition, and the time needed to complete the task was recorded with a stopwatch to the nearest 0.01 s.
Changes in five times sit to stand test | Baseline to 4-5 weeks after surgery
  Patients were instructed to perform the Five Times Sit to Stand Test (5STS) on a standardized armless chair (i.e., seating height between 41-45 cm, no elbow rests and wheels). After the cue "ready, set, go!", patients started the STS repetitions as rapidly as possible from the sitting position with their buttocks touching the chair to the full standing position, with their arms crossed over the chest. The 5STS test finished when the patients sit on the chair after the fifth repetition, and the time needed to complete the task was recorded with a stopwatch to the nearest 0.01 s.

CONTACTS AND LOCATIONS:
Locations (1):
- Portuguese Oncology Institute of Coimbra, Coimbra, Portugal